CLINICAL TRIAL: NCT03125811
Title: Value of Ondansetron Medication vs Inhaled Isopropyl Therapy in the Emergency Department (VOMIITED)
Acronym: VOMIITED
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Scott Crawford, Associate Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E17005
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Nausea; Vomiting
Keywords: Isopropyl alcohol; Zofran; antiemetics
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ethanol; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled Isopropyl Alcohol (IPA) (Active Comparator): Inhaled Isopropyl Alcohol (alcohol prep pad)
  Interventions: Other: Inhaled Isopropyl Alcohol (IPA)
- Oral Dissolvable Tablet Zofran (OZ) (Other): 4 mg Oral Dissolvable Tablet Zofran (ondansetron)
  Interventions: Drug: Oral Dissolvable Tablet Zofran (ondansetron)

INTERVENTIONS:
Other: Inhaled Isopropyl Alcohol (IPA) — Three doses within 60 minutes. Doses will occur at 0 minutes, 30 minutes, and 60 minutes. Each dose consists of 3 inhalations of one IPA prep pad. A new prep pad is used at each dose.
  Other Names: IPA; alcohol prep pad
  Arms: Inhaled Isopropyl Alcohol (IPA)
Drug: Oral Dissolvable Tablet Zofran (ondansetron) — Single dose 4 mg tablet at 0 minutes.
  Other Names: OZ
  Arms: Oral Dissolvable Tablet Zofran (OZ)

SUMMARY:
This study will compare two different ways to relieve nausea and vomiting in the Emergency Department. The usual treatment for nausea/vomiting is a drug called Zofran, but new studies have suggested that smelling alcohol pads can also help to relieve nausea and vomiting.

DETAILED DESCRIPTION:
Emergency physicians commonly use medications to alleviate nausea and vomiting. The medication Ondansetron is used in the emergency department and after surgery for this purpose. Inhaled isopropyl alcohol has been successfully used to decrease nausea and vomiting after surgery. No trial has compared inhaled isopropyl alcohol to Ondansetron in a clinical trial.

The author proposes to prospectively investigate extension of the established antiemetic efficacy of inhaled isopropyl alcohol for undifferentiated nausea in Emergency Department patients to the 30-minute post-intervention point that has been reported to be the frequent juncture of symptom relief. By introducing prolonged intervention, and re-dosing of established benefit, into this research, the author aims to reproduce the sustained antiemetic efficacy of inhaled isopropyl alcohol for undifferentiated nausea as demonstrated for post-operative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years presenting to the emergency department complaining of current nausea with or without episodes of emesis beginning within the previous 24hrs

Exclusion Criteria:

* Patients with known allergy to isopropyl alcohol
* Patients outside of the defined age range
* Patients with an inability to inhale through the nares (including recent upper respiratory infection)
* Patients greater than 20 weeks estimated gestation
* Patients with past medical history of gastroparesis, or hemoptysis
* Patients who have taken an antiemetic medication in the past 48 hours
* Patients demonstrating hemodynamic instability with systolic blood pressure <90 or tachycardia >120 bpm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Nausea Severity | 60 minutes
  Patient's nausea severity will be assessed at three time points by the study personnel using a verbal nausea rating scale over the course 60 minutes. Severity is scored 0-10 (0 = no nausea; 10 = severe nausea). Time points are at 0 minutes, 30 minutes, and 60 minutes.

SECONDARY OUTCOMES:
Emesis Event | 60 minutes
  Total number of emesis will be recorded for the 60 minute participation.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Crawford, MD, Principal Investigator — Texas Tech Universtiy Health Sciences Center El Paso
Locations (2):
- United States (2):
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - University Medical Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Myer PA, Mannalithara A, Singh G, Singh G, Pasricha PJ, Ladabaum U. Clinical and economic burden of emergency department visits due to gastrointestinal diseases in the United States. Am J Gastroenterol. 2013 Sep;108(9):1496-507. doi: 10.1038/ajg.2013.199. Epub 2013 Jul 16. PMID 23857475
- [Background] Braude D, Soliz T, Crandall C, Hendey G, Andrews J, Weichenthal L. Antiemetics in the ED: a randomized controlled trial comparing 3 common agents. Am J Emerg Med. 2006 Mar;24(2):177-82. doi: 10.1016/j.ajem.2005.08.017. PMID 16490647
- [Background] Patanwala AE, Amini R, Hays DP, Rosen P. Antiemetic therapy for nausea and vomiting in the emergency department. J Emerg Med. 2010 Sep;39(3):330-6. doi: 10.1016/j.jemermed.2009.08.060. Epub 2009 Dec 21. PMID 20022195
- [Background] Barrett TW, DiPersio DM, Jenkins CA, Jack M, McCoin NS, Storrow AB, Singleton LM, Lee P, Zhou C, Slovis CM. A randomized, placebo-controlled trial of ondansetron, metoclopramide, and promethazine in adults. Am J Emerg Med. 2011 Mar;29(3):247-55. doi: 10.1016/j.ajem.2009.09.028. Epub 2010 Mar 26. PMID 20825792
- [Background] Furyk JS, Meek RA, Egerton-Warburton D. Drugs for the treatment of nausea and vomiting in adults in the emergency department setting. Cochrane Database Syst Rev. 2015 Sep 28;2015(9):CD010106. doi: 10.1002/14651858.CD010106.pub2. PMID 26411330
- [Background] Ohashi Y, Nakai Y, Ikeoka H, Koshimo H, Esaki Y, Horiguchi S, Teramoto K, Nakaseko H. An experimental study on the respiratory toxicity of isopropyl alcohol. J Appl Toxicol. 1988 Feb;8(1):67-71. doi: 10.1002/jat.2550080111. PMID 3356866
- [Background] Gill MW, Burleigh-Flayer HD, Strother DE, Masten LW, McKee RH, Tyler TR, Gardiner TH. Isopropanol: acute vapor inhalation neurotoxicity study in rats. J Appl Toxicol. 1995 Mar-Apr;15(2):77-84. doi: 10.1002/jat.2550150204. PMID 7782562
- [Background] Winston AW, Rinehart RS, Riley GP, Vacchiano CA, Pellegrini JE. Comparison of inhaled isopropyl alcohol and intravenous ondansetron for treatment of postoperative nausea. AANA J. 2003 Apr;71(2):127-32. PMID 12776641
- [Background] Pellegrini J, DeLoge J, Bennett J, Kelly J. Comparison of inhalation of isopropyl alcohol vs promethazine in the treatment of postoperative nausea and vomiting (PONV) in patients identified as at high risk for developing PONV. AANA J. 2009 Aug;77(4):293-9. PMID 19731848
- [Background] Hines S, Steels E, Chang A, Gibbons K. Aromatherapy for treatment of postoperative nausea and vomiting. Cochrane Database Syst Rev. 2012 Apr 18;(4):CD007598. doi: 10.1002/14651858.CD007598.pub2. PMID 22513952
- [Background] Beadle KL, Helbling AR, Love SL, April MD, Hunter CJ. Isopropyl Alcohol Nasal Inhalation for Nausea in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2016 Jul;68(1):1-9.e1. doi: 10.1016/j.annemergmed.2015.09.031. Epub 2015 Dec 8. PMID 26679977